CLINICAL TRIAL: NCT01480167
Title: Prospective Randomized Investigation of Radiofrequency Targeted Vertebral Augmentation (The PRIORi-T Trial)
Brief Title: The PRIORi-T Trial--Prospective Randomized Investigation of Radiofrequency Targeted Vertebral Augmentation
Acronym: PRIORi-T
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: DFINE Inc. (Industry)
Responsible Party: Sponsor
Organization: Merit Medical Systems, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC-10-005 - PRIORI-T
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Painful Osteoporotic Vertebral Compression Fractures (VCF)
Keywords: VCF; Osteoporosis; Minimally Invasive; Non-operative management; Medical Management
MeSH Terms: conditions — Osteoporosis | interventions — Kyphoplasty; Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RF-TVA with STABILIT Vertebral Augmentation System (Active Comparator): All RadioFrequency-Targeted Vertebral Augmentation (RF-TVA) arm participants will be treated with the StabiliT Vertebral Augmentation System. This system is a commercially available device in the United States designed to perform percutaneous vertebral augmentation (also known as kyphoplasty).
  Interventions: Device: Vertebral Augmentation (STABILIT)
- Non Operative Management (Active Comparator): All non-operative management (NOM) arm participants will receive non-operative standard of care management, which can include: analgesics, bed rest, back braces, physiotherapy, rehabilitation programs, and walking aids according to standard practices of participating institutions.
  Interventions: Other: Non-operative Management

INTERVENTIONS:
Device: Vertebral Augmentation (STABILIT) — Vertebral Augmentation with the STABILIT Vertebral Augmentation System
  Other Names: Kyphoplasty; Radiofrequency Targeted Vertebral Augmentation (RF-TVA); Radiofrequency Kyphoplasty (RFK)
  Arms: RF-TVA with STABILIT Vertebral Augmentation System
Other: Non-operative Management — Conservative Care
  Other Names: Medical Management
  Arms: Non Operative Management

SUMMARY:
The objective of this post market clinical investigation is to evaluate the clinical effectiveness of a minimally invasive vertebral augmentation procedure, Radiofrequency-Targeted Vertebral Augmentation (RF-TVA) as compared to non-operative management (NOM) for the treatment of appropriately diagnosed acute (≤ 8 weeks) painful osteoporotic vertebral compression fractures (VCF).

DETAILED DESCRIPTION:
This is a multi-center, prospective, randomized, post marketing clinical trial designed to evaluate the clinical effectiveness of a minimally invasive procedure, Radiofrequency-Targeted Vertebral Augmentation (RF-TVA), compared to Non Operative Management (NOM) for the treatment of appropriately diagnosed, acute (≤ 8 weeks), painful, osteoporotic vertebral compression fractures. Eligible subjects will be randomly allocated to receive either RF-TVA or NOM in a 1:1 randomization ratio. Subjects will be followed for 12 months post procedure. Primary effectiveness will be determined by comparing the Visual Analogue Scale for each treatment group for back pain from the baseline to the 1-month post procedure visit and between treatment groups at 1-month.

Up to 15 sites will participate in this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 21 and ≤ 90 years of age.
2. Subject has one (1) to three (3) painful vertebral compression fracture(s) at T5-L5 due to primary or secondary osteoporosis (i.e. non-malignant) and recent history of sudden onset of pain in area of index vertebra (e).
3. Subject's index vertebra (e) is confirmed as the active source of back pain as evidenced by concordant pain and bone marrow edema via magnetic resonance imaging (MRI) or Computerized Tomography (CT) plus bone scan.
4. Subject has a history of vertebral fracture-related back pain ≤ 8 weeks old at time of enrollment (confirmed by medical history).
5. Subject has a pain related VAS score ≥ 5 on a scale of 0 to 10 at time of enrollment. Pain represents the worst level of back pain while standing, walking or elevating from chair, bed, or car during the preceding 24 hours associated with the index vertebra (e).
6. Subject has a Roland Morris Disability Questionnaire (RDQ) score ≥ 10 on scale of 0 to 24 at time of enrollment.
7. Subject is a suitable candidate for minimally invasive VCF procedure.
8. Subject has sufficient mental and physical capacity to comply with the Investigational Plan requirements and is willing and able to provide informed consent; agrees to release medical information for the purposes of this study; and agrees to comply with the Investigational Plan requirements and return for specified follow-up evaluations.
9. Subject is a male; a documented infertile female (either postmenopausal or surgical contraception); or is a non-pregnant, non-lactating female of childbearing potential who agrees to use a medically accepted method of birth control throughout the duration of the trial.

Exclusion Criteria:

1. Subject's VCF morphology is deemed unsuitable for RF-TVA in the judgment of the Investigator.
2. Subject requires additional non-kyphoplasty or vertebroplasty surgical treatment for the index fracture.
3. Subject has surgery to the spine planned for at least one (1) month following enrollment.
4. Subject has high-energy trauma-related and/or, non-osteoporotic vertebral fractures.
5. Subject has a spinal cord compression or significant canal compromise requiring decompression, in the judgment of the investigator.
6. Subject has a neurologic deficit associated with the vertebral level(s) to be treated that is more severe than radiculopathy (e.g. myelopathy, cauda equina syndrome).
7. Subject has irreversible coagulopathy or bleeding disorder.
8. Subject requires, at time of enrollment, the use of high-dose steroids (e.g. ≥ 100 mg prednisone or 20 mg dexamethasone per day), intravenous (IV) pain medication, or nerve block to control chronic back pain unrelated to index VCF(s).
9. Subject has significant clinical co-morbidities that may potentially interfere with the collection of data concerning pain and function.
10. Subject has a known allergy to device materials (e.g. polymethylmethacrylate (PMMA) or barium).
11. Subject has a contraindication to local or general anesthesia.
12. Subject has a medical and/or surgical condition contrary to the kyphoplasty or vertebroplasty procedure (e.g. presence of local or systemic infection).
13. Subject is receiving Worker's Compensation.
14. Subject is a prisoner.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement in back pain from baseline at the 1 month follow-up visit as measured by the Visual Analog Scale. | 1 month

SECONDARY OUTCOMES:
Change in VAS from baseline at the 3, 6, and 12 month follow-up visits. | 3, 6, and 12 months
Change in Roland-Morris Questionnaire (RDQ) from baseline at the 1, 3, 6, and 12 month follow-up visits. | 1,3,6,12 months
Change in SF-36 physical component score from baseline at the 1, 3, 6, and 12 month follow-up visits. | 1,3,6,12 months
Change in IOF Quality of Life Questionnaire from baseline at the 1, 3, 6, and 12 month follow-up visits. | 1,3,6,12 months

CONTACTS AND LOCATIONS:
Overall Officials: Allan Brook, M.D., Principal Investigator — Montefiore Hospital/Einstein Medical School
Locations (6):
- United States (6):
  - Washington University - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Department of Radiology, Lebanon, New Hampshire
  - Winthrop University Hospital, Department of Radiology, Mineola, New York
  - Montefiore Hospital/Einstein Medical School, Department of Radiology, The Bronx, New York
  - Penn State Hershey Medical Center, Department of Radiology, Hershey, Pennsylvania
  - Swedish Neuroscience Institute, Cherry Hill Campus, Department of Neurosurgery, Seattle, Washington